CLINICAL TRIAL: NCT02226094
Title: A Prospective, Randomized, Controlled Clinical Feasibility Investigation of the Safety and Efficacy of Deep Wave Trabeculoplasty (DWT) in Primary Open Angle Glaucoma (POAG) and Ocular Hypertension (OHT) Subjects
Brief Title: Safety and Efficacy of Deep Wave Trabeculoplasty (DWT) in Primary Open Angle Glaucoma and Ocular Hypertension
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: OcuTherix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DWT CIP 002
Record Dates: First submitted 2014-08-20; First posted 2014-08-27 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Primary Open-angle Glaucoma (POAG); Ocular Hypertension (OHT)
Keywords: intra-ocular pressure; primary open-angle glaucoma; intra ocular pressure; primary open angle glaucoma; glaucoma; deep wave trabeculoplasty; ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- DWT device dose A (Experimental): Deep Wave Trabeculoplasty (DWT) dose A (10 second spot treatments).
  Interventions: Device: DWT device dose A
- Ellex Tango SLT machine (Active Comparator): Selective Laser Trabeculoplasty (SLT)
  Interventions: Device: Ellex Tango SLT machine
- DWT Sham (Sham Comparator): Deep Wave Trabeculoplasty (DWT) but device not applied to ocular surface.
  Interventions: Device: DWT sham
- DWT device dose B (Experimental): Deep Wave Trabeculoplasty (DWT) dose B (20 second spot treatments).
  Interventions: Device: DWT device dose B

INTERVENTIONS:
Device: DWT device dose A — Deep Wave Trabeculoplasty (DWT) is an investigational device intended to reduce IOP in patients with POAG or OHT. The DWT device applies focal mechanical oscillation (low amplitude, sonic frequency) to the surface of the eye proximate the limbal region and anterior to the trabecular meshwork (TM). Mechanical oscillation of the TM by the DWT device is believed to initiate a physiological cascade to restore function of the TM, increase the outflow of aqueous humor and thereby decrease the IOP. DWT involves 24 spot treatments applied around the limbal region on the ocular surface. Dose A refers to 10 second spot treatments.
  Arms: DWT device dose A
Device: Ellex Tango SLT machine — Laser trabeculoplasty is the application of a laser beam to burn areas of the trabecular meshwork, located near the base of the iris, to increase fluid outflow. Selective laser trabeculoplasty (SLT) uses a Nd:YAG laser to target specific cells within the trabecular meshwork and create thermal damage.
  Arms: Ellex Tango SLT machine
Device: DWT device dose B — Same as DWT device dose A except 20 second spot treatments.
  Arms: DWT device dose B
Device: DWT sham — Same as DWT device dose A except device not applied to ocular surface.
  Arms: DWT Sham

SUMMARY:
The primary purpose of this study is to investigate the safety and efficacy of bilateral DWT in subjects with POAG or OHT compared to active and sham controls. The secondary purpose of the study is to investigate the durability, repeatability, and does response of the same.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 years or older.
* Subjects diagnosed with either POAG or OHT in both eyes. The diagnosis of POAG must include evidence of:

  1. Optic disc or retinal nerve fiber layer structural abnormalities (substantiated by OCT); and/or
  2. Visual field abnormality (substantiated with the Humphrey automated perimeter using the SITA Standard 24-2 testing algorithm. Mean deviation (MD) score must be -15dB < MD < 0dB.
* Subjects with a 9:00AM (+/- 1 hour) median IOP in both eyes that is:

  1. Greater than or equal to 18mmHg at the Screening Visit or have documented history of IOP being greater than or equal to 22mmHg;
  2. Greater than or equal to 22mmHg at both Eligibility Visits.
* Subjects currently using one or more topical medications to control their IOP.
* Subjects able and willing to comply with the protocol, including randomization assignment and all follow-up visits.
* Subjects that sign the informed consent form.

Exclusion Criteria:

* Subjects who are pregnant, lactating, or planning to become pregnant during the course of the study.
* Subjects with any form of glaucoma other than primary open-angle glaucoma (e.g., pseudo exfoliation or pigmentary glaucoma).
* Other exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percent decrease in IOP and change in dependence on IOP-lowering medications from baseline | 6 months
Intra-procedural and post-procedural adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Siy Uy, MD, Principal Investigator — Pacific Eye and Laser Institute; Edgar U. Leuenberger, MD, Principal Investigator — Asian Eye Institute; Maria I Yap-Veloso, MD, Principal Investigator — Asian Eye Institute
Locations (2):
- Philippines (2):
  - Asian Eye Institute, Makati City
  - Pacific Eye and Laser Institute, Makati City